CLINICAL TRIAL: NCT05682196
Title: Open-label, Randomized Controlled Trial to Assess Efficacy and Safety of Rituximab in Patients With Acute Rheumatic Fever in Africa
Brief Title: Rituximab in Patients With Acute Rheumatic Fever
Acronym: AGRAF-2
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: ethical controversy
Sponsor: African Academy of Methodology and Statistics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGRAF-2
Record Dates: First submitted 2022-12-15; First posted 2023-01-12 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Rheumatic Heart Disease in Children
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab plus standard of care (RTX) (Experimental): Rituximab i.v of two perfusions (375 mg/m²) administered in a 14 day-interval added to a standard of care treatment
  Interventions: Drug: Rituximab added to standard of care treatment
- Standard of care treatment (Control) (Active Comparator): Standard of care treatment
  Interventions: Drug: standard of care treatment alone

INTERVENTIONS:
Drug: Rituximab added to standard of care treatment — Rituximab with standard of care treatment
  Other Names: Rituximab with standard of care treatment
  Arms: Rituximab plus standard of care (RTX)
Drug: standard of care treatment alone — Standard of care treatment alone
  Arms: Standard of care treatment (Control)

SUMMARY:
Acute Rheumatic Fever is an autoimmune inflammatory post-infectious syndrome, mainly caused by type A streptococcus. It is characterized as an inadequate immune response. It may provoke carditis, combined with articular, skin and neurologic signs. Only carditis, prevalent in 60% of acute rheumatic diseases, may provoke valvular sequels, which define rheumatic cardiopathy. Antibiotherapy based on penicillin is the standard treatment of both acute rheumatic fever and its prevention. Although no anti-inflammatory treatment has proved its efficacy, with or without steroids anti-inflammatory treatments are administered in acute episode of ARF. Up to date, only prevention strategies have shown efficacy.

DETAILED DESCRIPTION:
Acute Rheumatic Fever is an autoimmune inflammatory post-infectious syndrome, mainly caused by type A streptococcus. It is characterized as an inadequate immune response. It may provoke carditis (which associates valvular leakages, cardiac conduction system troubles, and pericardial signs), combined with articular, skin and neurologic signs. Only carditis, prevalent in 60% of acute rheumatic diseases, may provoke valvular sequels, which define rheumatic cardiopathy. Prevalence of acute rheumatic disease (ARD) in pproximately 6 cases per 1000 children in Sub-Saharan Africa countries, whereas prevalence in developed countries is less than a case per 100 000 children, with an annual incidence of 470 000 cases and almost 230 000 deaths annually worldwide. Carditis affect between 15 and 20 million people worldwide, mostly children and young adults from low and middle-income countries. This prevalence may be underestimated. In 2007, our team conducted a study in Mozambique and Cambodia that highlighted that, through a screening based on systematic echocardiography in children from several schools, approximately 2/3 of them had asymptomatic and unknown cardiac lesions, which cannot be screened only with a clinical examination. Role of B-type lymphocytes (B cells) in auto-immune diseases physiopathology is nowadays largely accepted and justifies, in certain auto-immune diseases, the use of therapeutics that target and destroy B cells. Rituximab is a CD-20-specific monoclonal chimeric antibody, indicated to treat B lymphomas, where its efficacy and safety have changed the management of these diseases. Recently, it is thought to use Rituximab in auto-immune diseases. Antibiotherapy based on penicillin is the standard treatment of both acute rheumatic fever and its prevention. Although no anti-inflammatory treatment has proved its efficacy, with or without steroids anti-inflammatory treatments are administered in acute episode of ARF. Up to date, only prevention strategies have shown efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between >= 5 and < 17 years old;
* Diagnosed acute rheumatic fever with at least one progressive rheumatic valvular lesion confirmed through a cardiac echography.
* Informed consent, signed and dated by both parents or legal guardians of the patient

Exclusion Criteria:

* Simultaneous active infection, such as HIV, hepatitis B, C, tuberculosis, Epstein-Barr virus (EBV), or history of frequent, unusual or serious infections ;
* Pathologies likely to affect immunity (cancer, multiple sclerosis, diabetes, other auto-immune diseases)
* Recent history of drug administration that may affect the immune system, for the past 4 weeks (immunosuppressive drugs, corticosteroids, anticancer drugs);
* Hypersensitivity reaction to rituximab or one of its components. Hypersensitivity to penicillin
* History of monoclonal antibodies administration
* Recent vaccination (less than a month) or planned within the 12 months after randomization;
* History of heart failure
* Renal failure with a creatinine clearance <45 ml/min/1,73m²
* Pregnancy (a negative urinary test is necessary for women who had their first menstruations or aged 14 years old and more)
* Patients diagnosed with Guillain-Barré syndrome
* Patient with at least one of the following biological features : Hemoglobin < 8,5 g/dL, Platelets < 100 G/L, Neutrophils < 1,5 G/L, Leucocytes < 3 G/L, AST or ALT increased > 2,5 the normal superior limit)
* Any acute or chronic infection clinically significant which would limitate the patient's capacity to follow up the study protocol, which remains under appreciation of the investigator.
* Any participation in another clinical trial in the 6 months before the pre-randomization visit

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Rheumatic valvular lesions rate | 6 months post randomization
  Rheumatic valvular lesions rate, measured by echocardiography

SECONDARY OUTCOMES:
Incidence of rheumatic valvular lesions | 14 days, 3, 6 and 12 months post-randomization
  Rate of rheumatic valvular lesions will be compared between groups
Serious adverse events rates | at 14 days, 3, 6, and 12 months after randomization
  Serious adverse events rate will be compared between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Fann Hospital, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided